CLINICAL TRIAL: NCT02364934
Title: Effect of Different Anesthetics on Pharmacokinetics and Pharmacodynamics of Rocuronium in Closed-Loop Muscle Relaxant Infusion System
Brief Title: Pharmacokinetics and Pharmacodynamics of Rocuronium in Closed-Loop Infusion System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Donglai Yan, Chief, Tianjin Medical University General Hospital
Other Study IDs: IRB014-090-01
Record Dates: First submitted 2014-12-23; First posted 2015-02-18 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: TOF; Sex
Keywords: rocuronium; sex; elderly; Close-loop infusion system
MeSH Terms: conditions — Coitus | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Propofol: Propofol is intravenously administrated during anesthesia maintenance in patients (18-65 years old)
  Interventions: Drug: Propofol
- Sevoflurane: Sevoflurane (inhalation) is administrated during anesthesia maintenance in patients (18-65 years old)
  Interventions: Drug: Sevoflurane
- Propofol (elderly): Propofol is intravenously administrated during anesthesia maintenance in patients (≥65 years old)
  Interventions: Drug: Propofol
- Sevoflurane (elderly): Sevoflurane (inhalation) is administrated during anesthesia maintenance in patients (≥65 years old)
  Interventions: Drug: Sevoflurane
- Propofol (men): Propofol is intravenously administrated during anesthesia maintenance in men (18-65 years old)
  Interventions: Drug: Propofol
- Sevoflurane (men): Sevoflurane (inhalation) is administrated during anesthesia maintenance in men (18-65 years old)
  Interventions: Drug: Sevoflurane
- Propofol (women): Propofol is intravenously administrated during anesthesia maintenance in women (18-65 years old)
  Interventions: Drug: Propofol
- Sevoflurane (women): Sevoflurane (inhalation) is administrated during anesthesia maintenance in women (18-65 years old)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — This study was designed to determine the dose requirements for rocuronium, administered by continuous infusion to maintain a stable 90-99% T1 depression (depression of the first twitch in the train-of-four, TOF) in adult, elderly and different sex patients under sufentanil and propoful anaesthesia.
  Groups: Propofol; Propofol (elderly); Propofol (men); Propofol (women)
Drug: Sevoflurane — This study was designed to determine the dose requirements for rocuronium, administered by continuous infusion to maintain a stable 90-99% T1 depression (depression of the first twitch in the train-of-four, TOF) in adult, elderly and different sex patients under sufentanil and sevoflurane anaesthesia.
  Groups: Sevoflurane; Sevoflurane (elderly); Sevoflurane (men); Sevoflurane (women)

SUMMARY:
To explore and compare the effects of propoful, sevoflurane, and a combination of both on the pharmacokinetics and pharmacodynamics of rocuronium.

To discover and confirm sex differences on the pharmacokinetics and pharmacodynamics of rocuronium.

To evaluate and examine aged people on the pharmacokinetics and pharmacodynamics of rocuronium.

DETAILED DESCRIPTION:
Rocuronium is a non-depolarizing neuromuscular blocking agent with intermediate duration of action and without significant cumulative properties, suitable for continuous infusion. This study was designed to determine the dose requirements for rocuronium, administered by continuous infusion to maintain a stable 90-99% T1 depression (depression of the first twitch in the train-of-four, TOF) in adult, elderly and different sex patients under sufentanil and propoful, sevoflurane, or propoful + sevoflurane anaesthesia.

Methods Two hundred and ten patients, ASA physical status group I and II undergoing elective surgical procedures were studied. Pateients with neuromuscular and metabolic diseases, morbid obesity or receiving medication known to influence neuromuscular transmission were excluded from the study.

Anaesthesia Patients will be assigned at random to receive propofuol, sevolurane or propoful+sevoflurane anaesthesia. All patients will induced with midazolam, 0.1 mg/kg, sufentnail, 0.5 μg/kg, etomidate, 0.3 mg/kg and rocuronium, 0.6 mg/kg. In the propoful group, anaesthesia will be continued with propoful and sufentanil. The doseage of propotul and sufentanil will be adjusted by the blood pressure and heart rate of the patients. In the sevoflurane group, anaesthesia will be continued with sevoflurane (2%) and sufentanil. The doseage of sufentanil will be adjusted by the blood pressure and heart rate of the patients. The doseage of propoful and sufentanil will be adjusted by the blood pressure and heart rate of the patients.

Heart rate, invasive blood pressure, pulse and core body temperature were monitored throughout the procedure. The core body temperature was main tained between 36°C and 37°C using a warming blanket. Positive pressure ventilation was used to maintain the end-tidal CO2 between 4.5 kPa and 5.5 kPa. The inspired and end-tidal concentrations of carbon dioxide and volatile anaesthestics were monitored by a multigas monitor.

Neuromuscular transmission was monitored by recording the electromyographic (EMG) activity of the adductor pollicis muscle resulting from the supra- maximal stimulation of the ulnar nerve with train-of- four (TOF), 2 Hz for 2 s, applied at 10-s intervals. The ulnar nerve was stimulated through surface electrodes applied at the wrist, using square-wave currents of 0.2 ms duration. Ten minutes were allowed for the stabilization of anaesthesia and the EMG tracing before the intubating dose of rocuronium, 0.6 mg/kg, was given by the anaesthesiologist.

Rocuronium infusion A personal computer, working in a closed-loop system with the Relaxograph and a syringe infusion pump was used to administer rocuronium at the rate necessary for a stable 90-99% block of the first twitch response (1%<T1<10%). The infusion of rocuronium was started automatically when T1 returned to 5% of the control value. The initial infusion rate was set at 10 mg/kg/min, and subsequently adjusted by the computer. Every 10 s the computer received data (T1 value) from the Relaxograph. If T1 increased above 10%, the infusion rate was increased by 2/3. If T1 increased above 15%, a bolus dose (0.06 mg/kg) was administered automatically to avoid an undesirable return of the muscle strength during surgery. The neuromuscular block was considered stable if T1 changed by no more than 2% over a 10-min observation period. The rocuronium infusion was automatically stopped if three consecutive T1 values equalled 0. The working mode (automatic or manual), the last six T1 values and the 15-min T1 trend could be observed on screen. The anaesthesiologist could override the computer-set infusion rate at any time, by changing the working mode from automatic to manual, and stop the infusion when the surgery was completed.

All neuromuscular transmission data, as well as the data on the infusion rate during the closed-loop system feed-back infusion of the relaxant, were saved in a Microsoft Excel compatible computer file.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status group I and II
* elective surgical procedures
* The subject has given written informed consent to participate

Exclusion Criteria:

* Coronary heart disease, bronchial asthma, cardiac, lung, hepatic and renal insufficiency
* Severe HBP, obesity (BMI>30)
* Neuromuscular and metabolic diseases
* Receiving medication known to influence neuromuscular transmission
* Pregnancy, psychiatric disease
* Allergy history
* Inability to understand the Study Information Sheet and provide a written consent to take part in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA physical status group I and II undergoing elective surgical procedures were studied. Pateients with neuromuscular and metabolic diseases, morbid obesity or receiving medication known to influence neuromuscular transmission were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Time to give additional rocuromium | 24h
  A personal computer, working in a closed-loop system with the Relaxograph and a syringe infusion pump was used to administer rocuronium at the rate necessary for a stable 90-99% block of the first twitch response (1%<T1<10%).

SECONDARY OUTCOMES:
Total dose of rocuronium | 24h
  A personal computer, working in a closed-loop system with the Relaxograph and a syringe infusion pump was used to administer rocuronium at the rate necessary for a stable 90-99% block of the first twitch response (1%<T1<10%).
Bispectral index（BIS） | 24h
  The test is measured by bispectral index（BIS）form the patient arrive the operation room to leave the operation room.
Time to spontaneous breathing recovery, eye opening, extubation | 24h
  Time to spontaneous breathing recovery, eye opening, extubation
Agitation score | 24h
  The test is measured after extubation, 5min、10min and 15min after arrival at PACU